CLINICAL TRIAL: NCT05961748
Title: Registry of Multicenter Brain-Heart Comorbidity in China
Acronym: BHC-C
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xiaolin Chen, MD, Director, Beijing Tiantan Hospital
Other Study IDs: KY2022-221-02
Record Dates: First submitted 2023-07-07; First posted 2023-07-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Heart Disease; Cardiac Arrest; Atrial Fibrillation; Heart Failure; Aortic Diseases; Subarachnoid Hemorrhage; Intracerebral Hemorrhage; Cerebral Infarction; Occlusion and Stenosis of Precerebral Arteries; Occlusion and Stenosis of Cerebellar Arteries; Cerebral Aneurysm; Moyamoya Disease; Arteriovenous Malformation of Cerebral Vessels
MeSH Terms: conditions — Myocardial Ischemia; Heart Arrest; Atrial Fibrillation; Heart Failure; Aortic Diseases; Subarachnoid Hemorrhage; Cerebral Hemorrhage; Cerebral Infarction; Bites and Stings; Intracranial Aneurysm; Moyamoya Disease; Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multi-disciplinary assessment — Multi-disciplinary assessment

SUMMARY:
This study is a multi-center, prospective, registry study. This research was supported by the National Key Research and Development Program. To establish a domestic multi-center, large-scale "brain-heart comorbidity" dynamic database platform including clinical, sample database, image and other multi-dimensional information requirements, through the construction of a multi-center intelligent scientific research integration platform based on artificial intelligence.

Any of newly diagnosed cardiovascular related diseases were identified via ICD-10-CM codes: I21, I22, I24 (Ischaemic heart diseases) [i.e., ACS], I46 (cardiac arrest), I48 (Atrial fibrillation/flutter), I50 (Heart failure), I71 (Aortic disease), I60 (subarachnoid hemorrhage), I61 (intracerebral hemorrhage), I63 (Cerebral infarction), I65 (Occlusion and stenosis of precerebral arteries), I66 (Occlusion and stenosis of cerebral arteries), I67.1 (cerebral aneurysm), I67.5 (moyamoya diseases), Q28.2 (Arteriovenous malformation of cerebral vessels).

The data is stored on the brain-heart comorbidity warehouse via a physical server at the institution's data centre or a virtual hosted appliance. The brain-heart comorbidity platform comprises of a series of these appliances connected into a multicenter network. This network can broadcast queries to each appliance. Results are subsequently collected and aggregated. Once the data is sent to the network, it is mapped to a standard and controlled set of clinical terminologies and undergoes a data quality assessment including 'data cleaning' that rejects records which do not meet the brain-heart comorbidity quality standards. The brain-heart comorbidity warehouse performs internal and extensive data quality assessment with every refresh based on conformance, completeness, and plausibility (http://10.100.101.65:30080/login).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* Any of newly diagnosed cardiovascular-related diseases were identified via ICD-10-CM codes: I21, I22, I24 (Ischaemic heart diseases) [i.e., ACS], I46 (cardiac arrest), I48 (Atrial fibrillation/flutter), I50 (Heart failure), I71 (Aortic disease), I60 (subarachnoid hemorrhage), I61 (intracerebral hemorrhage), I63 (Cerebral infarction), I65 (Occlusion and stenosis of precerebral arteries), I66 (Occlusion and stenosis of cerebral arteries), I67.1 (cerebral aneurysm), I67.5 (moyamoya diseases), Q28.2 (Arteriovenous malformation of cerebral vessels).

Exclusion Criteria:

·refuse to participate in the registry

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * age > 18 years old
  * Any of newly diagnosed cardiovascular-related diseases were identified via ICD-10-CM codes: I21, I22, I24 (Ischaemic heart diseases) [i.e., ACS], I46 (cardiac arrest), I48 (Atrial fibrillation/flutter), I50 (Heart failure), I71 (Aortic disease), I60 (subarachnoid hemorrhage), I61 (intracerebral hemorrhage), I63 (Cerebral infarction), I65 (Occlusion and stenosis of precerebral arteries), I66 (Occlusion and stenosis of cerebral arteries), I67.1 (cerebral aneurysm), I67.5 (moyamoya diseases), Q28.2 (Arteriovenous malformation of cerebral vessels).
  Exclusion Criteria:
  ·refuse to participate in the registry
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Participants with Composite of All-Cause Mortality and Cardiovascular Outcomes | At discharge/30 days
  The occurrence of all-cause mortality, coronary artery disease event, stroke (ischemic or hemorrhagic), heart failure, or atrial fibrillation etc.
All-Cause Mortality | At discharge/30 days
  The occurrence of death
Rate of Participants with Composite of Cardiovascular Outcomes | At discharge/30 days
  The occurrence of coronary artery disease event, stroke (ischemic or hemorrhagic), heart failure, or atrial fibrillation etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, MD, Study Chair — Beijing Tiantan Hospital; Yong Cao, MD, Study Director — Beijing Tiantan Hospital; Dong Xu, MD, Principal Investigator — Beijing Tiantan Hospital; Zening Jin, MD, Principal Investigator — Beijing Tiantan Hospital; Hao Wang, MD, Principal Investigator — Beijing Tiantan Hospital; Shuai Kang, MD, Principal Investigator — Beijing Tiantan Hospital; Yu Chen, MD, Principal Investigator — Beijing Tiantan Hospital; Qingyuan Liu, MD, Principal Investigator — Beijing Tiantan Hospital; Runting Li, MD, Principal Investigator — Beijing Tiantan Hospital; Heze Han, MD, Principal Investigator — Beijing Tiantan Hospital; Wenxiong Song, MD, Principal Investigator — Beijing Tiantan Hospital; Jionghao Xue, MD, Principal Investigator — Beijing Tiantan Hospital; Minghao Liu, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (14):
- China (14):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Shenzhen Qianhai Shekou Free Trade Zone Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Shanxi, Shanxi
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan